CLINICAL TRIAL: NCT06612151
Title: A Multicenter, Randomized, Controlled, Open-label, Phase III Study to Compare the Efficacy and Safety of YL201 Versus Topotecan Hydrochloride in Subjects with Relapsed Small Cell Lung Cancer
Brief Title: A Phase III Study of YL201 in Relapsed Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: MediLink Therapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YL201-CN-302-01
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-09

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Topotecan; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- YL201 (Experimental): Participants are randomized to receive YL201 monotherapy intravenously on Day 1 of each 3-week cycle at RP3D dose level, until progressive disease (PD), unacceptable toxicity, or withdrawal of consent as specified in the protocol.
  Interventions: Drug: YL201
- topotecan hydrochloride for injection (Active Comparator): Participants are randomized to receive topotecan hydrochloride intravenously, on Days 1 to 5 of each 3-week cycle per prescribing information, until PD, unacceptable toxicity, or withdrawal of consent as specified in the protocol.
  Interventions: Drug: topotecan hydrochloride for injection

INTERVENTIONS:
Drug: YL201 — Patients will be treated with YL201 intravenous (IV) infusion once every 3 weeks (Q3W) as a cycle at RP3D dose level.
  Arms: YL201
Drug: topotecan hydrochloride for injection — Topotecan hydrochloride will be administered intravenously per prescribing information.
  Arms: topotecan hydrochloride for injection

SUMMARY:
This study was designed to compare the efficacy and safety of YL201 with Topotecan Hydrochloride in subjects with relapsed small cell lung cancer (SCLC).

DETAILED DESCRIPTION:
The primary objective of this study is to assess whether treatment with YL201 prolongs overall survival (OS) compared with treatment of topotecan hydrochloride among subjects with relapsed SCLC.

The secondary objectives of the study are to further evaluate the efficacy, safety, pharmacokinetics, and immunogenicity of YL201, and the correlation between B7-H3 expression level and the efficacy of YL201.

ELIGIBILITY:
Inclusion Criteria:

1. Sign and date the informed consent form prior to the start of any study-specific qualification procedures.
2. Aged ≥18 and ≤75 years, male or female.
3. ECOG PS 0 or 1.
4. Life expectancy ≥ 3 months.
5. Histologically or cytologically confirmed SCLC. Subjects with combined SCLC or any transformed SCLC are not eligible.
6. Has limited-stage or extensive-stage disease at study entry, with progression on or after first-line platinum-based therapy (at least 2 cycles).
7. At least one measurable lesion according to RECIST version 1.1.
8. Subjects are willing to provide tumor tissue (freshly obtained or archived) for detection of B7-H3 expression.
9. Adequate organ function.

Exclusion Criteria:

1. History of other malignant tumors within 5 years prior to the first dose of study drug. Subjects cured by radical treatment are not included, such as basal cell carcinoma, squamous cell carcinoma of skin, superficial bladder cancer, carcinoma in situ of the cervix, or breast cancer in situ.
2. Previously received B7-H3-targeted therapy, including antibody, antibody-drug conjugate (ADC), and chimeric antigen receptor T cell (CAR-T).
3. Previously received treatment with a topoisomerase I inhibitor or an ADC consisting of a topoisomerase I inhibitor.
4. Inadequate washout period for prior anti-tumor treatment before the first dose of study drug.
5. Received systemic steroids or other immunosuppressive therapy within 2 weeks before the first dose of study drug.
6. Received any live vaccine within 4 weeks before the first dose of study drug or intend to receive a live vaccine during the study.
7. Presence of brain stem or meningeal metastases, spinal cord metastases or compression.
8. Presence of central nervous system (CNS) metastasis. Participants with treated brain metastases are eligible if the metastases are asymptomatic and stable, and no immediate local or systemic treatment is needed within 2 weeks before the first dose.
9. Presence of pleural effusion, pericardial effusion, or ascites with clinical symptoms or requiring repeated drainage.
10. Has an uncontrolled concurrent disease.
11. Presence of severe uncontrolled cardiovascular disorder.
12. History of interstitial lung disease (ILD) or pneumonitis that required corticosteroids, or current ILD/pneumonitis
13. Concomitant pulmonary disorder leading to clinically severe respiratory impairment.
14. Chronic autoimmune or inflammatory diseases requiring or receiving systemic therapy within 2 years prior to the first dose.
15. Serious infections within 4 weeks prior to the first dose.
16. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
17. Unresolved toxicities from previous antitumor therapy.
18. Known hypersensitivity to any component of any study drug; history of severe allergy or known history of serious hypersensitivity to other monoclonal antibodies or recombinant protein products, or history of severe infusion reactions.
19. Pregnancy, breastfeeding, or women planning to become pregnant or breastfeed during the study.
20. Any illness, medical condition, organ system dysfunction, or social situation deemed by the investigator to be likely to interfere with a subject's ability to sign informed consent, adversely affect the subject's ability to cooperate and participate in the study, or compromise the interpretation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
To compare the OS of YL201 versus topotecan hydrochloride in subjects with relapsed SCLC. | Approximately within 36 months
  (OS) defined as the time interval from the first randomization to death due to any cause.

SECONDARY OUTCOMES:
To compare Investigator-assessed progression-free survival (PFS) of YL201 versus topotecan hydrochloride in subjects with relapsed SCLC. | Approximately within 36 months
  PFS defined as the time interval from randomization to the first documented PD or death due to any cause, whichever occurs first.
To compare Investigator-assessed objective response rate (ORR) of YL201 versus topotecan hydrochloride in subjects with relapsed SCLC. | Approximately within 36 months
  ORR defined as the proportion of subjects who achieve a best overall response (BOR) of complete response (CR) or partial response (PR).
To compare duration of response (DoR) as assessed by the investigator of YL201 versus topotecan hydrochloride in subjects with relapsed SCLC. | Approximately within 36 months
  DoR defined as the time interval from the first documentation of response (CR or PR) to the first documentation of PD or death, whichever occurred first.
To compare time to response (TTR) as assessed by the investigator of YL201 versus topotecan hydrochloride in subjects with relapsed SCLC. | Approximately within 36 months
  TTR defined as the time interval from randomization to the first documentation of response (CR or PR).
To compare disease control rate (DCR) assessed by the investigator of YL201 versus topotecan hydrochloride in subjects with relapsed SCLC. | Approximately within 36 months
  DCR defined as the proportion of subjects with a BOR of CR, PR, or stable disease (SD).
To evaluate the incidence and severity of adverse events (AEs) of YL201. | Approximately within 36 months
  AEs are assessed based on NCI CTCAE v5.0.
To evaluate the concentration-time data for YL201, total antibody, and payload | Approximately within 36 months
To characterize the PK parameter AUC | Approximately within 36 months
Characterize the PK parameter Cmax | Approximately within 36 months
To characterize the PK parameter Ctrough | Approximately within 36 months
To characterize the PK parameter CL | approximately within 36 months
Characterize the PK parameter Vd | approximately within 36 months
Characterize the PK parameter t1/2 | Approximately within 36 months
Assessment of B7H3 expression level in tumor tissue and the correlation between the expression level and the efficacy of YL201. | Approximately within 36 months
Assessment of the number of subjects who are Anti-Drug Antibody (ADA)-positive at any time and who have a treatment-emergent ADA | Approximately within 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No